CLINICAL TRIAL: NCT05344066
Title: MIDDAS-GDM: A Two-Arm Randomised Feasibility Protocol Trial of an Intermittent Low-Energy Diet (ILED) in Women With Gestational Diabetes and Obesity in Greater Manchester
Brief Title: Manchester Intermittent Diet in Gestational Diabetes Acceptability Study
Acronym: MIDDAS-GDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B01410
Record Dates: First submitted 2022-02-11; First posted 2022-04-25 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2023-12

CONDITIONS: Gestational Diabetes; Gestational Diabetes Mellitus in Pregnancy; Intermittent Fasting; Pregnancy Related; Diabetes; Diabetes in Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Intermittent Fasting; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomised two-arm feasibility trial
Masking Description: Non blinded (statistician and laboratory staff will remain blinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best NHS Care (Active Comparator): Best National Health Service (NHS) Care
  Interventions: Other: Best NHS Care
- Intermittent Low Energy Diet (Experimental): Intermittent Low Energy Diet
  Interventions: Other: Intermittent Low Energy Diet

INTERVENTIONS:
Other: Best NHS Care — Personalised advice and support from a diabetes dietician to follow NICE healthy eating diet and physical activity recommendations for GDM.
  Arms: Best NHS Care
Other: Intermittent Low Energy Diet — Two non-consecutive days of a food based 1000 kcal diet and five days of the NICE healthy eating diet and physical activity recommendations for the best NHS care group.
  Arms: Intermittent Low Energy Diet

SUMMARY:
A two-arm non-blinded randomised feasibility protocol trial designed to assess the feasibility, safety, and acceptability of an intermittent low energy diet (ILED) vs best National Health Service (NHS) care in women with gestational diabetes and obesity in Greater Manchester.

DETAILED DESCRIPTION:
Overall aim:

The aim of this trial is to test the safety, feasibility, and acceptability of an ILED in GDM to inform a future large-scale RCT.

Background:

Up to 16% of pregnant women in the United Kingdom develop GDM with rising rates due to increasing rates of obesity and maternal age. GDM affects both maternal and neonatal outcomes and is a high burden to patients and the NHS through frequent clinic visits, monitoring, and costly medications such as insulin. The National Institute for Health and Care Excellence (NICE) guidelines advocate healthy diet (with increased physical activity [PA]) as first-line therapy for GDM with approximately 30% progressing to metformin and/or insulin treatment. Our Patient and Public Involvement and Engagement work demonstrates that women with GDM are keen for alternative dietary interventions to reduce their need for medications. It has been shown that intermittent low energy diets improve glycaemic control in type-2 diabetes. The investigators wish to test the utility of ILED in GDM.

Primary Aim: to test the safety, feasibility, and acceptability of an ILED in GDM to inform a future large-scale RCT.

Primary Objectives:

* Uptake rate
* Recruitment rate
* Retention rate
* Adherence to the dietary interventions
* Completion of self-assessed glucose and ketone readings

Safety outcomes:

* Percentage of women following ILED/best NHS care with hypoglycaemia (episodes of blood glucose of <3.0mmol/mol)
* Percentage of women who develop significant ketonaemia in both groups (defined as ≥1.0mmol/L)
* Percentage of neonatal hypoglycaemic episodes requiring intervention, neonatal birth weight, gestational age at delivery, hyperbilirubinaemia/jaundice, and/or admission to Special Care Baby Unit or neonatal intensive care, and stillbirths
* The incidence and rate of other adverse events (e.g. headaches, lethargy, constipation, or complications requiring hospital admission) between the start of the trial intervention and delivery.

Secondary outcomes

* Completeness of collection of trial endpoints
* Fidelity of delivery of the interventions
* Qualitative analysis of the acceptability and implementation of the interventions

Exploratory outcomes The following outcomes will be explored without statistical inference.

1. Maternal outcomes:

   * The percentage of women requiring metformin and/or insulin
   * Four-point capillary glucose profiles during third trimester
   * Change in fasting blood test results between baseline measurements, 36-37 weeks' gestation, and 12 weeks post-delivery
   * Mode of delivery, development of preeclampsia, polyhydramnios (maximum liquor volume pool depth ≥8 cm)
   * Quality of life and health status questionnaires (WHOQoL-BREF and SF-36 questionnaires)
2. Foetal outcomes:

   * Foetal weight
   * Gestational age at delivery

Method:

We aim to recruit 48 women with GDM diagnosed between 24-30 weeks gestation from antenatal clinics at Wythenshawe and St Mary's hospitals, Manchester Foundation Trust, over 13 months starting in November 2022. Participants will be randomised (1:1) to ILED (2 low-energy diet days/week of 1000kcal and 5 days/week of the best NHS care healthy diet and physical activity advice) or best NHS care 7 days/week until delivery of their baby. Primary outcomes include uptake and retention of participants to the trial, and adherence to both dietary interventions. Safety outcomes will include birthweight, gestational age at delivery, neonatal hypoglycaemic episodes requiring intervention, neonatal hyperbilirubinaemia, admission to special care baby unit or neonatal intensive care unit, stillbirths, the percentage of women with hypoglycaemic episodes requiring third-party assistance, and significant maternal ketonaemia (defined as ≥1.0mmol/L) Secondary outcomes will assess the fidelity of delivery of the interventions, and qualitative analysis of participant and healthcare professionals' experiences of the diet. Exploratory outcomes include the number of women requiring metformin and/or insulin.

Qualitative evaluation:

Investigators will undertake qualitative analysis of the experiences and thoughts of approximately 5 participants per group and healthcare professionals delivering the interventions.

Anticipated impact and dissemination:

This study will inform the feasibility and design of a definitive RCT of ILED versus best NHS care in GDM. Findings will be disseminated to health professionals and patients through published articles, conference presentations and patient networks in collaboration with the patient and public involvement and engagement panel.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women ≥18 years
2. BMI of ≥27.5kg/m2 or a BMI ≥25 kg/m2 in high risk minority ethnic group (i.e. South Asian, Black African, African Caribbean) and <50 kg/m2 at booking appointment (8-12 weeks' gestation)
3. Newly diagnosed GDM according to local diagnostic criteria (fasting glucose ≥5.3mmol/l and/or 2-hour postprandial glucose ≥8.5mmol/l in a 75g OGTT) scheduled to receive first line diet and physical activity (best NHS care)
4. 24-30 weeks pregnant at screening appointment

Exclusion Criteria:

1. Pregestational type 1 or type 2 diabetes.
2. Fasting glucose of ≥7 or 2-hour postprandial of ≥11 on OGTT (immediate intervention with medication would be required in this group of women)
3. Current multiple pregnancy
4. Maturity Onset Diabetes of the Young (MODY)
5. Significant comorbid disease that in PI's opinion would preclude participation in the study e.g. chronic kidney disease, significant cardiac disease, history of disordered eating or severe psychological problems.
6. Current participation in a GDM medication treatment trial
7. People who are not capable of providing informed consent or adhering to the monitoring and safety protocols
8. People who have previously had bariatric surgery for weight loss including gastric bypass and sleeve gastrectomy, and/or those prescribed weight loss medications (e.g. orlistat).
9. Medications at the time of the OGTT that may interfere with results (e.g. high dose oral steroids, immunosuppressants)
10. Previous history of intrauterine growth restriction
11. Women who have lost more than 5% of their weight from booking appointment to screening appointment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Trial recruitment rate | Duration of trial (68 weeks)
  Uptake to trial will be measured as a percentage of eligible participants who consent to participate in the trial per month.
Retention to the trial | Duration of trial (68 weeks)
  Retention rate will be measured as the percentage of participants who complete all scheduled 8 visits.
Trial uptake | Duration of trial (68 weeks)
  Trial uptake will be measured as the percentage of eligible participants who consent to participate in the trial.
Adherence to the interventional intermittent low-calorie diet over course of study | From randomisation (at 24-30 weeks' gestation) to delivery.
  Self-reported adherence to the two potential low-calorie days per week expressed as a percentage of the potential low-calorie days in the intermittent low energy diet group.
Adherence to capillary glucose and ketone measurements over course of study | From randomisation (at 24-30 weeks' gestation) to delivery
  The number of self-assessed glucose (4 times a day) and ketone (3 times a day on two days of the week) measurements in both groups over the course of the study.
Episodes of hypoglycaemia requiring intervention | From 24-30 weeks' gestation until delivery.
  The percentage of women with self-reported hypoglycaemia (capillary blood glucose of <3.0 mmol/l) will be measured and compared between groups.
Episodes of ketonaemia requiring intervention | From 24-30 weeks' gestation until delivery.
  The percentage of women with self-reported significant ketonaemia (capillary ketones >1 mmol/l) will be measured and compared between groups.
Rates of neonatal hyperbilirubinaemia/jaundice | From delivery until final visit at 12-13 weeks' postpartum
  Percentage of neonatal hyperbilirubinaemia/jaundice (defined as a total serum bilirubin level above 86 μmol/l) episodes will be recorded in both groups.
Rates of neonatal hypoglycaemia | From delivery until 12 hours post-delivery
  Percentage of neonatal hypoglycaemic episodes requiring intervention (blood glucose checked 2-hours post delivery and 2-hours thereafter for 12 hours) will be recorded in both groups.
Neonatal birthweight | At delivery
  Neonatal birth weight will be measured in kilograms and recorded in both groups.
Neonatal gestational age at delivery | At delivery
  Gestational age at delivery will be measured in weeks and recorded in both groups.
Gestational age at delivery | At delivery
  Gestational age at delivery in weeks will be recorded in both groups.
Rates of admission to special care baby unit or neonatal intensive care | From delivery until final visit at 12-13 weeks' postpartum
  Rates of admission to Special Care Baby Unit or Neonatal Intensive Care will be recorded in both groups.
Number of stillbirths | At delivery
  Number of stillbirths will be recorded in both groups.

SECONDARY OUTCOMES:
Number of completed scheduled patient contacts | Duration of trial (68 weeks)
  Completion of scheduled patient contacts with the trial dietitian and gestational diabetes midwife will be recorded and compared between groups.
Completion rates of food diaries | 4 day food diaries at 24-30 weeks' gestation, 34-35 weeks' gestation, 36-37 weeks' gestation, and 12-13 weeks postpartum.
  Participants will be asked to complete 4-day food diaries for 4 weeks of the trial at 24-28 weeks' gestation, 34-35 weeks' gestation, 36-37 weeks' gestation, and 12-13 weeks postpartum. They will also be given the option of recording diaries during the other weeks as this may help with their adherence. Completion rates of the food diaries each week across the whole intervention as a percentage of weeks in both groups will inform the utility of food diaries for tracking diet behaviour in both groups
Completion rates of International Physical Activity Questionnaire (IPAQ) | IPAQ questionnaire at 24-30 weeks' gestation, 34-35 weeks' gestation, 36-37 weeks' gestation, and 12-13 weeks postpartum.
  Participants will be asked to complete the IPAQ during 4 weeks of the trial at 24-28 weeks' gestation, 34-35 weeks' gestation, 36-37 weeks' gestation, and 12-13 weeks postpartum. Completion rates will be measured as a percentage of weeks completed in both groups.
The acceptability of the dietary interventions will be explored qualitatively | 12-13 weeks' postpartum
  A subset of participants in both groups (approximately 5 participants from each group) will be invited to an optional qualitative substudy which will involve one semi-structured interview at the end of the intervention. Participants will be asked about their experiences and thoughts regarding the intervention. Key themes will be identified using Braun and Clarke's thematic analysis to identify key issues around the acceptability of the test intervention.

OTHER OUTCOMES:
Percentage of participants commencing metformin | From 24-30 weeks' gestation until delivery.
  The percentage of women commencing metformin will be measured.
Percentage of participants commencing insulin | From 24-30 weeks' gestation until delivery.
  The percentage of women commencing insulin will be measured.
Changes in HbA1c (mmol/mol) | Recorded at 24-30 weeks' gestation, 36-37 weeks' gestation, and at 12-13 weeks postpartum
  Bloods will be taken at 27-29 weeks' gestation, 36-37 weeks' gestation, and at 12-13 weeks postpartum. Changes in HbA1c between these time points will be compared within and between groups and expressed in mmol/mol.
Changes in fasting glucose (mmol/L) | Recorded at 24-30 weeks' gestation, 36-37 weeks' gestation, and at 12-13 weeks postpartum
  Bloods will be taken at 27-29 weeks' gestation, 36-37 weeks' gestation, and at 12-13 weeks postpartum. Changes in fasting glucose between these time points will be compared within and between groups and expressed in mmol/L.
Changes in fasting insulin (mU/L) | Recorded at 24-30 weeks' gestation, 36-37 weeks' gestation, and at 12-13 weeks postpartum
  Bloods will be taken at 27-29 weeks' gestation, 36-37 weeks' gestation, and at 12-13 weeks postpartum. Changes in insulin levels between these time points within and between groups will be compared and expressed in mU/L.
Oral Glucose Tolerance Test (mmol/L) result | 11-13 weeks' postpartum
  Oral Glucose Tolerance Test (OGTT) will be completed at 11-13 weeks postpartum. Fasting and 2 hour postprandial bloods will be measured and the percentage of women with a diagnosis of residual diabetes according to the World Health Organization (WHO) criteria will be reported in both groups.
Changes in the value of Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | Recorded at 24-30 weeks' gestation, 36-37 weeks' gestation, and at 12-13 weeks postpartum
  HOMA-IR will be calculated from fasting glucose and insulin measurements [(fasting insulin mU/L x fasting glucose nmol/L)/22.5] assessed at 27-29 weeks' gestation, 36-37 weeks' gestation, and at 12-13 weeks postpartum. Changes in HOMA-IR between these time points will be compared within and between groups.
Changes in maternal health status | Recorded at 24-30 weeks' gestation, 31-33 weeks' gestation, 36-37 weeks' gestation, and at 12-13 weeks postpartum
  Health status (SF-36) questionnaires will be completed in both groups and scores compared both within and between groups. Scores range from 1-100; the lower the score the more the disability, the higher the score the more favourable the health state.
Changes in maternal quality of life | Recorded at 24-30 weeks' gestation, 31-33 weeks' gestation, 36-37 weeks' gestation, and at 12-13 weeks postpartum
  Quality of life (WHOQoL-BREF) questionnaires will be completed in both groups and scores compared both within and between groups. This questionnaire measures four domains (physical health, psychological, social relationships and environment). Final scores range between 1-100; higher scores indicate a higher quality of life.
Changes in maternal glycaemic control | From 24-30 weeks' gestation until delivery
  Four-point capillary glucose profiles (four times daily) between 27-29 weeks' gestation and delivery will be compared within and between groups. The percentage of women within target ranges will be reported within and between groups (fasting <5.3 and 1 hour postprandial <7.8 mmol/l).
Mode of delivery | At delivery
  Mode of delivery will be recorded in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Basil Issa, Principal Investigator — Manchester Foundation Trust
Locations (1):
- Manchester University NHS Foundation trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient identifiable data will not be shared.
  Anonymised trial data will be available on reasonable request to the investigators.
Time Frame: Data will be available following data analysis and publication, and will be accessible for 5-10 years.
Access Criteria: To be confirmed

REFERENCES:
- [Derived] Dapre E, Issa BG, Harvie M, Su TL, McMillan B, Pilkington A, Hanna F, Vyas A, Mackie S, Yates J, Evans B, Mubita W, Lombardelli C. Manchester Intermittent Diet in Gestational Diabetes Acceptability Study (MIDDAS-GDM): a two-arm randomised feasibility protocol trial of an intermittent low-energy diet (ILED) in women with gestational diabetes and obesity in Greater Manchester. BMJ Open. 2024 Feb 10;14(2):e078264. doi: 10.1136/bmjopen-2023-078264. PMID 38341207